CLINICAL TRIAL: NCT03793348
Title: A Prospective, Multi-center, Pivotal Study to Evaluate the Safety and Efficacy of the Cytrellis Micro-Coring Device for the Treatment of Moderate to Severe Facial Wrinkles
Brief Title: Study to Evaluate the Safety and Efficacy of the Cytrellis Micro-Coring Device for the Treatment of Moderate to Severe Facial Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS 700-00052
Record Dates: First submitted 2018-12-18; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Wrinkle
Keywords: facial wrinkles; skin laxity; sagging skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Micro-exisional skin removal (Experimental): Micro-coring of skin on the facial and neck areas will be conducted in one treatment and followed for 90 days post treatment.
  Interventions: Device: MCD

INTERVENTIONS:
Device: MCD — Micro coring skin removal with automated coring device

SUMMARY:
Study evaluating the efficacy of a micro coring device for the treatment of moderate to severe check wrinkles

DETAILED DESCRIPTION:
Up to 35 subjects who meet the inclusion/exclusion criteria will be treated. All subjects will be monitored for a period of 90 days post treatment.

Study results will be assessed with the following:

* Lemperle Scale
* Investigator GAIS Scale
* Subject Satisfaction Scale

ELIGIBILITY:
Inclusion Criteria:

* Males and females 40-70 years of age
* Fitzpatrick Skin Type I to IV as judged by the Investigator
* Cheek areas are at least a score of 3 using the Lemperle Wrinkle Assessment Scale as judged by the Investigator
* Able to provide written informed consent, understand and willing to comply with all study related procedures and follow-up visits.

Exclusion Criteria:

* Lesions suspicious for any malignancy or the presence of actinic keratosis, melasma, vitiligo, cutaneous papules/nodules or active inflammatory lesions in the areas to be treated
* History of keloid formation or hypertrophic scarring
* History of trauma or surgery to the treatment areas in the past 6 months
* Scar present in the areas to be treated
* Silicone injections in the areas to be treated
* Injection of dermal fillers, fat or botulinum toxin, as well as any minimally invasive/invasive medical device for skin treatment, in the study treatment areas, within the past 6 months (i.e., dermabrasion, laser, RF devices)
* Active smokers (0.5 pack/day) or having quit within 3 months prior to treatment
* Active, chronic, or recurrent infection
* History of compromised immune system or currently being treated with immunosuppressive agents
* History of sensitivity to analgesic agents, Aquaphor®, topical or local anesthetics (e.g., lidocaine, benzocaine, procaine) or chlorhexidine, povidone-iodine or epinephrine
* Excessive sun exposure and use of tanning beds or tanning creams within 30 days prior to treatment
* Treatment with aspirin or other blood thinning agents within 14 days prior to treatment
* History or presence of any clinically significant bleeding disorder
* Any issue that, at the discretion of the Investigator, would interfere with assessment of safety or efficacy or compromise the subject's ability to participate in the study
* Treatment with an investigational device or agent within 30 days before treatment or during the study period

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-08-21 (Estimated)

PRIMARY OUTCOMES:
Assess level of wrinkle improvement using the Lemperle Wrinkle Severity Scale | 90 day post treatment
  A mean change of 1 point or greater reduction in cheek wrinkle severity at 90 days post treatment using the Lemperle Wrinkle Severity Scale, as assessed by (3) blinded Independent Reviewers Lemperle Scale:
  No wrinkles =0 Just perceptible wrinkles =1 Shallow wrinkles=2 Moderately deep wrinkles=3 Deep wrinkles, well-defined edges =4 Very deep wrinkles, redundant fold=5

SECONDARY OUTCOMES:
Assess aesthetic improvement using Global Aesthetic Improvement Scale | 90 day post treatment
  Overall aesthetic improvement level per Principal Investigator at 90 days compared to baseline on the Global Aesthetic Improvement Scale.
  Very Much Improved (Optimal cosmetic result)=3 Much Improved (Marked improvement from the initial condition, but not completely optimal)=2 No Change (The appearance is essentially the same as baseline)=0 Worse (The appearance is worse than the original condition)= -1 Much Worse (Marked worsening in appearance from the initial condition)= - 2 Very Much Worse (Obvious worsening in appearance from the initial condition)=- 3
Assess aesthetic improvement using Subject Satisfaction Scale | 90 day post treatment
  Satisfaction with the aesthetic appearance of the treatment area per Subject Satisfaction Scale compared to baseline.
  Extremely dissatisfied=0 Somewhat dissatisfied=1 Slightly dissatisfied=2 Neither satisfied or dissatisfied=3 Slightly satisfied=4 Somewhat satisfied=5 Extremely satisfied=6
Assess aesthetic improvement in wrinkles using OCT images (optional) | Baseline to Day 90 post treatment
  Assessment of improvement using OCT images with Vista software to determine wrinkle depth reduction, comparing pre-treatment depth to post treatment depth.
Assess efficacy results using Canfield Software,, by comparing the changes in wrinkles at baseline and 90 days post treatment. | Baseline to Day 90 post treatment
  Validated Canfield software comparing baseline wrinkles to day 90 follow up wrinkles via automated photo analysis.
Assess safety profile by recording of adverse events | Adverse events will be recorded immediately treatment, Day 1, Day 7, Day 30, Day 60 and Day 90 post treatment. Ad hoc assessment can occur upon subject report of AE.
  The incidence and severity of systemic and local adverse events will be recorded by the PI at all visits and a 14 day diary completed by each subject will also be collected.
Assess safety profile by reviewing completed 14 day subject diary for potential side effects. | For 14 days post treatment
  14 day diary completed by each subject will record potential side effects, level of severity (mild = 1; moderate = 2; severe = 3), and end date of the potential side effects.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Miami Dermatology & Laser Institute, Miami, Florida
  - Laser and Skin Surgery of New York, New York, New York
  - The Office of Brian Biesman, M.D., Nashville, Tennessee
  - Dallas Plastic Surgery Institute, Dallas, Texas